CLINICAL TRIAL: NCT01271530
Title: The Impact of an Arm Ergometry Training Programme on Cardiovascular Fitness, Energy Cost of Walking and Fatigue in Prior Polio Patients
Brief Title: Arm Cycling to Improve Fitness in Polio Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Post Polio Support Group Ireland (Unknown); Beaumont Hospital (Other)
Responsible Party: Principal Investigator, Deirdre Murray, Clinical Specialist Physiotehrapist in Neurosciences and PhD student, Royal College of Surgeons, Ireland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RoyalCSI DMurray
Record Dates: First submitted 2010-12-10; First posted 2011-01-06 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Postpoliomyelitis Syndrome
Keywords: Late Effects of Polio; Cardiovascular Fitness; Fatigue; Energy cost of Walking; Pain
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Fatigue; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Upper Limb Ergometry
- Control (No Intervention)

INTERVENTIONS:
Other: Upper Limb Ergometry — Cardiovascular training will be performed using upper limb ergometers at home for 8 weeks. Each subject will receive an individually prescribed programme and will begin exercising for at least ten minutes per day three days per week. If an individual has difficulty exercising for 10 minutes continuously, the 10 minute session may be broken into 2-3 minute bursts of exercise, with one minute rests. Subjects will aim to increase exercise durations to 20 minutes per day five days per week and will exercise at moderate to high intensities.
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effect of upper limb cardiovascular training on fitness, energy cost of walking, fatigue and pain in polio survivors. Polio survivors often have difficulty accessing aerobic forms of exercise due to limitations in mobility, pain associated with walking and fatigue. This can result in becoming physically unfit and places polio survivors at risk of secondary heath problems due to inactivity. A large percentage of polio survivors have lower limb involvement but have strong arms. The participants in this study will exercise at home using simple arm cycles for 8 weeks. They will attend for assessment on two occasions. All exercise will be prescribed by a Physiotherapist and includes measures to ensure safety while exercising at home.

DETAILED DESCRIPTION:
The American College of Sports Medicine (ACSM) recommendations state that stable muscle groups should be utilised for exercise in polio survivors and that patients with severe atrophic polio or with recent weakness should not exercise, while March of Dimes (2001) recommend not exercising muscle groups where new weakness is being experienced. Floor or treadmill walking or lower limb cycling may also aggravate pain in those with lower limb weakness and altered lower limb biomechanics.

Training with an upper limb ergometer is likely to be an appropriate form of exercise in patients with good, stable upper limb strength. One small, but well designed, trial of upper limb ergometry over 16 weeks resulted in a 19% increase in maximal oxygen uptake (VO2max) in 10 postpolio subjects exercising 3 times per week (Kriz et al 1992). ACSM recommend using a Schwinn Air-DyneTM four limb exerciser; however this is an expensive and bulky piece of equipment and is unlikely to be feasible for ongoing use by community dwelling polio survivors.

A small upper limb ergometer may be a cost effective, accessible option for exercise for community dwelling polio survivors. A closely monitored and carefully prescribed cardiovascular fitness programme may enable polio survivors, who have gained control of symptoms of fatigue and pain through changes in lifestyle and activity, to increase fitness and perhaps subsequently reduce energy cost of walking.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed history of Poliomyelitis affecting at least one lower limb, confirmed by the consultant Neurologist, Beaumont Hospital, Dublin, and documented in the medical chart.
* Capable of walking for 6 minutes, with or without an aid or appliance (as reported by the patient).
* Good upper limb strength, confirmed objectively by Quantitative Muscle Analysis (QMA) (Maximum Voluntary Isometric Contraction (MVIC)). MVIC scores of 7 out of 10 tested upper limb movements must lie above the 5th percentile of the normal range.
* Completion of the Physical Activity Readiness Questionnaire (PAR-Q) and cleared by medical practitioner as safe for exercise if indicated.
* Aged > 18 and < 75 NOTE: Participants must be resident in Ireland.

Exclusion Criteria:

* History of unstable cardiac or respiratory conditions
* Uncontrolled hypertension
* Oxygen dependence
* Significant upper limb pain (Visual Analogue Scale > 4 or more than 3 specific sites of pain)
* Severe fatigue (Fatigue Severity Scale > 5)
* Recent onset of upper limb weakness or severe upper limb weakness (< 5th percentile on more than 3 tested upper limb movements, either reported by the patient or measured using Quantitative Muscle assessment.
* Steroid use in last 3 months
* Use of medications which may influence cardiovascular testing (Beta-blockers etc)
* Pregnant Women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Six Minute Arm Test | Eight weeks
  The Six Minute Arm test is a submaximal cardiovascular fitness test. The American College of Sports Medicine recommend submaximal fitness testing, limited to 6-12 minutes and using either four limb ergometry or an upper limb ergometer in prior polio patients. The 6 Minute Arm Test (Hol et al 2007) is such a submaximal upper limb exercise test, which has been developed and found valid and reliable in spinal cord injury.
The Physical Activity Scale for Persons with Physical Disabilities | Eight weeks
  The Physical Activity Scale for Persons with Physical Disabilities is a subjectively reported survey of activity levels in people with physical disabilities. Preliminary validation has been completed by Washburn et al (2002).

SECONDARY OUTCOMES:
Upper Limb Maximal Voluntary Isometric Contraction | Eight weeks
  Upper limb strength will be measured to determine suitability for exercise and to measure any training related changes. Maximal voluntary isometric contraction of the upper limbs will be measured using fixed dynamometry with the Quantitative Muscle Analysis system. Shoulder abduction, adduction, elbow flexion and extension and hand grip will be measured.
Body Mass Index and Waist to hip Ratio | Eight weeks
  Body composition will be assessed using Body Mass Index and Waist to hip ratio will be used to measure risk due to overweight / obesity.
Hand Grip Motor Fatigue | Eight weeks
  Hand grip motor fatigue will be measured using Quantitative Muscle Analysis. This will be measured pre and post training to provide an indication of changes in motor fatigue occurring with training.
Short Form 36 Version 2 (SF-36 v2) | Eight weeks
  The SF-36v2 is a tool developed by Ware (www.sf-36.org), which measures health status. It has been used previously in polio survivors (Vasiliadis et al 2002, Gonzales et al 2006)
Short Form McGill Pain Questionnaire version 2 (SF-MPQ-2) | Eight weeks
  Pain will be assessed using the SF-MPQ-2. The SF-MPQ-2 questionnaire is a well-developed tool for quantitative assessment of pain (Dworkin et al 2009).
Physiological Cost Index | Eight weeks
  The Physiological Cost Index is a measure, which aims to estimate energy cost of walking, using walking speed and change in heart rate from baseline.
The Fatigue Severity Scale | Eight weeks
  The Fatigue Severity Scale is a commonly used questionnaire used to assess subjective fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre E Murray, BSc, Principal Investigator — Royal College of Surgeons in Ireland; Dara Meldrum, MSc, Study Director — Royal College of Surgeons in Ireland; Frances Horgan, PhD, Study Director — Royal College of Surgeons in Ireland; Orla Hardiman, MD, Study Chair — Beaumont Hospital; Roisin Moloney, BSc, Study Director — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Derived] Murray D, Meldrum D, Moloney R, Campion A, Horgan F, Hardiman O. The effects of a home-based arm ergometry exercise programme on physical fitness, fatigue and activity in polio survivors: protocol for a randomised controlled trial. BMC Neurol. 2012 Dec 13;12:157. doi: 10.1186/1471-2377-12-157. PMID 23234560